CLINICAL TRIAL: NCT06077136
Title: Efficacy of Upper Limb Exercises Using Whole Body Vibration on Muscle Tone, Motor Skills, Handgrip Strength, and Quality of Life in Children With Spastic Upper Motor Neuron Lesion
Brief Title: Whole Body Vibration in Rehabilitation of Spastic Cerebral Palsy
Acronym: WBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, assistant professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2023-380
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: the model of this study will be 2 parallel arms where one arm will receive regular physical therapy including exercises to the upper limb and the experimental group will receive the same physical therapy plus upper limb exercises applied using the whole body vibration device
Who Masked: Outcomes Assessor
Masking Description: Concealed allocation will be performed by a researcher who will not be involved in the treatment or assessment. Permuted blocks will be used to ensure an equal 1:1 allocation ratio. Due to the nature of the study, the assessor and the data analyzer will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular physical therapy group (Active Comparator): this group will receive regular physical therapy 3 -5 times per week. this program will be designed according to the needs of each child. strength, stretch, facilitation, splinting, coordination, and functional exercises are examples of the components of the programs.
  Interventions: Other: standard physical therapy
- whole body vibration (Experimental): in addition to the regular exercises, selected arm exercises will be performed while the child is under whole-body vibration. using (Galileo® MED 25 TT, Germany; 2021 model) with the following parameters:
  * WBV session duration: 10 minutes (rest periods can be incorporated
  * frequency: 12 Hz
  * Amplitude: 2 (fixed)
  * duration of each exercise: 2-3 minutes
  Interventions: Other: whole body vibration; Other: standard physical therapy

INTERVENTIONS:
Other: whole body vibration — 3 sessions per week consisted of different types of exercises, all of which were performed while the child will be is under WBV using (Galileo® MED 25 TT, Germany; 2021 model) with the following parameters:
  * WBV session duration: 10 minutes (rest periods can be incorporated (1-2 minutes maximum 3 times during the session)
  * frequency: 12 Hz
  * Amplitude: 2 (fixed)
  * duration of each exercise: 2-3 minutes
  * starting positions differ according to each exercise; upper limb weight-bearing and weight shift (from prone, prone on elbows, sitting, standing).
  * upper limb active exercises using toys/ balls / wand. Involving throwing, catching, transfer between both hands (according to the abilities of each child).
  * coordination exercises by asking the child to approximate the index finger of both hands together, perform finger-to-nose (eyes open and closed), and finger-to-therapist finger exercises.
  Other Names: WBV
  Arms: whole body vibration
Other: standard physical therapy — all children will receive regular exercises according to their developmental abilities such as stretching, strengthening, facilitation, or inhibition as well as functional exercises. exercise sessions will be 3 times per week fo
  Other Names: exercises

SUMMARY:
Spasticity is one of the most common features in children with cerebral palsy (CP) and is evident in the majority of CP types such as hemiplegia, diplegia, quadriplegia, etc. Children with spastic upper motor neuron lesions often experience difficulties with muscle tone and movement, impacting their functional abilities and quality of life. Conventional treatments such as physical therapy and medication have demonstrated positive effects in the management of spasticity. However, alternative interventions like whole body vibration (WBV) have gained attention due to their potential to modulate muscle tone and improve functional outcomes. WBV involves the transmission of mechanical vibrations to the whole body or specific body parts. These vibrations stimulate sensory receptors and elicit muscular responses, potentially leading to improved muscle tone regulation and reduced spasticity.

DETAILED DESCRIPTION:
Several studies have investigated the effects of WBV on spasticity management. These studies have reported various outcomes, providing valuable insights into the potential benefits of this intervention. Previous studies showed an immediate reduction of spasticity of the calf muscle, increased the range of the popliteal angle, and improved step length, step width, foot angle, and walking speed.

The current study seeks to address some of the limitations observed in previous research. It employs a randomized controlled trial design with a predetermined sample size, enhancing the statistical power and generalizability of the findings. The intervention group will receive supervised upper limb exercises using WBV, while the control group will receive conventional therapy. By comparing these two groups, the study aims to provide more robust evidence regarding the specific effects of WBV on muscle tone and spasticity. Furthermore, the current study will utilize standardized assessment tools to measure muscle tone, spasticity, and functional outcomes pre-and post-intervention. This will allow for a comprehensive evaluation of the effects of WBV on spasticity management, encompassing both objective measures and functional improvements.

ELIGIBILITY:
Inclusion Criteria:

* age between 5 and 14 years,
* who had a diagnosed with spastic cerebral palsy by a pediatrician,
* 1-3 on Ashworth Scale (MAS) for upper limb muscles
* whose parents/guardians sign the informed consent,
* who were willing to complete the study.

Exclusion Criteria:

* Children with anatomical disorder or deformity in the upper limb,
* Children who received a botulinum toxin injection in the upper limb muscles during the last six months
* Surgery in the lower extremity during the previous year
* Severe associated neurological diseases as epilepsy
* Poor nutritional status.
* Those who do not agree to participate in the study.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth scale (MAS) for muscle tone | at baseline
  For clinical assessment of spasticity, the Modified Ashworth scale (MAS) will be used to assess the level of calf muscle spasticity. The assessor will apply passive ankle dorsiflexion on the affected side and determine the appropriate grade of spasticity. MAS grades range from 0, for normal muscle tone to 4 for extreme spasticity.
Modified Ashworth scale (MAS) for muscle tone | after the end of the treatment (after 4 weeks)
  For clinical assessment of spasticity, the Modified Ashworth scale (MAS) will be used to assess the level of calf muscle spasticity. The assessor will apply passive ankle dorsiflexion on the affected side and determine the appropriate grade of spasticity. MAS grades range from 0, for normal muscle tone to 4 for extreme spasticity.
APILHAND-Kids scale for fine motor skills | baseline
  ABILHAND-Kids is a parent-reported questionnaire measuring manual ability in children with cerebral palsy (CP). It includes 21 specific items. The Parent is asked to fill in the questionnaire by estimating their child's ease or difficulty in performing each activity by choosing "Impossible", "Difficult" or "Easy". The final score will be obtained using software available on http://rssandbox.iescagilly.be/ .
APILHAND-Kids scale for fine motor skills | after the end of the treatment (after 4 weeks)
  ABILHAND-Kids is a parent-reported questionnaire measuring manual ability in children with cerebral palsy (CP). It includes 21 specific items. The Parent is asked to fill in the questionnaire by estimating their child's ease or difficulty in performing each activity by choosing "Impossible", "Difficult" or "Easy". The final score will be obtained using software available on http://rssandbox.iescagilly.be/ .
eye-hand coordination using Mayro Device | at baseline
  using Mayro Device, Tyromotion, a device with a large touch screen that allows many training and assessment options. On the screen, multiple marks are arranged to form a circle with one mark located in the center. The child will be asked to trace these marks to make a final figure of a star. Errors will be calculated, and the final results will reflect the score of the child where higher score s means better achievement
eye-hand coordination using Mayro Device | after the end of the treatment (after 4 weeks)
  using Mayro Device, Tyromotion, a device with a large touch screen that allows many training and assessment options. On the screen, multiple marks are arranged to form a circle with one mark located in the center. The child will be asked to trace these marks to make a final figure of a star. Errors will be calculated, and the final results will reflect the score of the child where higher score s means better achievement
handgrip strength using Myro device | at baseline
  Using the ball (a specific accessory of the Mayro device) , the child will be asked to hold and squeeze the ball as hard as possible while the ball is attached to the Mayro device. The sensors within the ball will determine the pressure exerted by the child and the score will be recorded.
handgrip strength using Myro device | after the end of the treatment (after 4 weeks)
  Using the ball (a specific accessory of the Mayro device) , the child will be asked to hold and squeeze the ball as hard as possible while the ball is attached to the Mayro device. The sensors within the ball will determine the pressure exerted by the child and the score will be recorded.
The quality of life using paediatric Cerebral Palsy Quality of Life (CP QoL) questionnaire | at baseline
  Quality of life questionnaire covers the age ranges of 4-12 (i.e., CP QoL-Child). and 13-18 (i.e., CP QoL-Teen). Both CP QoL-Child and CP QoL-Teen were reported to be validated tools with strong psychometric properties and clinical utility. The translated Arabic version of CP-QOL questionnaire (caregiver form) is valid and reliable. the higher scores mean better QoL
The quality of life using paediatric Cerebral Palsy Quality of Life (CP QoL) questionnaire | after the end of the treatment (after 4 weeks)
  Quality of life questionnaire covers the age ranges of 4-12 (i.e., CP QoL-Child). and 13-18 (i.e., CP QoL-Teen). Both CP QoL-Child and CP QoL-Teen were reported to be validated tools with strong psychometric properties and clinical utility. The translated Arabic version of CP-QOL questionnaire (caregiver form) is valid and reliable. the higher scores mean better QoL

CONTACTS AND LOCATIONS:
Locations (1):
- Hisham Hussein, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No